CLINICAL TRIAL: NCT02196038
Title: REHAB-HF: A Trial of Rehabilitation Therapy in Older Acute Heart Failure Patients
Brief Title: A Trial of Rehabilitation Therapy in Older Acute Heart Failure Patients
Acronym: REHAB-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00028221; R01AG045551 (NIH)
Record Dates: First submitted 2014-07-15; First posted 2014-07-21 (Estimated); Results first posted 2021-06-23 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2020-09

CONDITIONS: Acute Decompensated Heart Failure
Keywords: heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attention Control (Other): Usual care group with bi-weekly contact from study staff
  Interventions: Behavioral: Attention Control
- multi-domain rehabilitation intervention (Active Comparator): Individual, tailored, progressive, physical function rehabilitation intervention
  Interventions: Behavioral: multi-domain rehabilitation intervention

INTERVENTIONS:
Behavioral: multi-domain rehabilitation intervention — Individual, tailored, progressive physical function rehabilitation intervention
  Arms: multi-domain rehabilitation intervention
Behavioral: Attention Control — Usual care with bi-weekly contact from study staff
  Arms: Attention Control

SUMMARY:
REHAB-HF: A Trial of Rehabilitation Therapy in Older Acute Heart Failure Patients, is a multicenter, randomized, attention-controlled, single-blind trial designed to examine the hypothesis that, in addition to standard care, a novel, tailored, progressive, multi-domain rehabilitation intervention administered to older patients with acute decompensated heart failure (ADHF) beginning early during hospitalization and continuing for 12 weeks will improve physical function and key clinical outcomes, including the rate of rehospitalization.

DETAILED DESCRIPTION:
There will be three lead centers, Wake Forest Baptist Health along with Thomas Jefferson University and Hospital-Co-Investigator Dr. David Whellan, and Duke University Medical Center-Co-Investigator Dr. Christopher O'Connor. Each center may recruit up to 3 geographically close, tightly affiliated 'satellite' sites under their management and budgetary control. Together, these sites will recruit a total of 352 consenting patients ≥ 60 years old hospitalized with ADHF. Following informed consent and baseline testing, the participants will be randomized in a 1:1 fashion to receive a 12-week novel, progressive, multi-domain rehabilitation and exercise training intervention or attention control. The multi-domain rehabilitation intervention will include endurance, mobility, strength, and balance training and will be tailored based on participant performance in each of these domains. It will begin upon randomization during the hospitalization and will continue 3 times per week in an outpatient setting. Participants randomized to the attention control arm will receive all services ordered by their primary physician and will be contacted bi-weekly by study staff. All participants will undergo measures of physical function and quality of life at baseline, 1 month, and 3 months. Clinical events will be monitored for 6 months following the index hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years old
* In the hospital setting >24 hours for the management of ADHF, or diagnosed with ADHF after being hospitalized for another reason. ADHF will be confirmed by the study physician, and will be defined according to the Food and Drug Administration definition of hospitalized heart failure as a combination of symptoms, signs, and HF-specific medical treatments.

Exclusion Criteria:

* Acute myocardial infarction
* Planned discharge other than to home or a facility where the participant will live independently
* Already actively participating in formal, facility-based cardiac rehabilitation

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2014-09; Primary Completion 2020-06-15 (Actual); Study Completion 2020-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dalane W. Kitzman, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (3):
- United States (3):
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Thomas Jefferson University and Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Damluji AA, Bruce SA, Reeves G, Pastva AM, Bertoni AG, Mentz RJ, Whellan DJ, Kitzman DW, deFilippi CR. Circulating Biomarkers as Predictors of Improvement in Physical Function in Hospitalized Older Adults With Geriatric Syndromes: Findings From the REHAB-HF Trial. Circ Heart Fail. 2026 Jan 7:e013251. doi: 10.1161/CIRCHEARTFAILURE.125.013251. Online ahead of print. PMID 41500239
- [Derived] Corsi DR, Dikdan S, Upadhyay N, Chen H, Kitzman DW, Mentz R, Whellan DJ, Frisch DR. Atrial Fibrillation Status and Physical Rehabilitation in Older Patients With Acute Decompensated Heart Failure: An Analysis From the REHAB-HF Trial. J Am Heart Assoc. 2024 Oct;13(19):e034366. doi: 10.1161/JAHA.124.034366. Epub 2024 Sep 18. PMID 39291487
- [Derived] Gilbert ON, Mentz RJ, Bertoni AG, Kitzman DW, Whellan DJ, Reeves GR, Duncan PW, Nelson MB, Blumer V, Chen H, Reed SD, Upadhya B, O'Connor CM, Pastva AM. Relationship of Race With Functional and Clinical Outcomes With the REHAB-HF Multidomain Physical Rehabilitation Intervention for Older Patients With Acute Heart Failure. J Am Heart Assoc. 2023 Nov 7;12(21):e030588. doi: 10.1161/JAHA.123.030588. Epub 2023 Oct 27. PMID 37889196
- [Derived] Pandey A, Kitzman DW, Nelson MB, Pastva AM, Duncan P, Whellan DJ, Mentz RJ, Chen H, Upadhya B, Reeves GR. Frailty and Effects of a Multidomain Physical Rehabilitation Intervention Among Older Patients Hospitalized for Acute Heart Failure: A Secondary Analysis of a Randomized Clinical Trial. JAMA Cardiol. 2023 Feb 1;8(2):167-176. doi: 10.1001/jamacardio.2022.4903. PMID 36598761
- [Derived] Nelson MB, Shiroma EJ, Kitzman DW, Duncan PW, Reeves GR, Whellan DJ, Mentz RJ, Chen H, Pastva AM. Physical activity and relationship to physical function, quality of life, and cognitive function in older patients with acute decompensated heart failure. Am Heart J. 2023 Feb;256:85-94. doi: 10.1016/j.ahj.2022.11.002. Epub 2022 Nov 11. PMID 36372251
- [Derived] Whellan D, McCarey MM, Chen H, Nelson MB, Pastva AM, Duncan P, Mentz RJ, Kitzman DW, Reeves G, Reed SD. Quality of Life Trajectory and Its Mediators in Older Patients With Acute Decompensated Heart Failure Receiving a Multi-Domain Rehabilitation Intervention: Results From the Rehabilitation Therapy in Older Acute Heart Failure Patients Trial. Circ Heart Fail. 2022 Dec;15(12):e009695. doi: 10.1161/CIRCHEARTFAILURE.122.009695. Epub 2022 Nov 8. PMID 36345825
- [Derived] Peters AE, Kitzman DW, Chen H, Nelson MB, Pastva AM, Duncan PW, Reeves GR, Upadhya B, Whellan DJ, Mentz RJ. Obesity Status and Physical Rehabilitation in Older Patients Hospitalized With Acute HF: Insights From REHAB-HF. JACC Heart Fail. 2022 Dec;10(12):918-927. doi: 10.1016/j.jchf.2022.07.008. Epub 2022 Sep 7. PMID 36164731
- [Derived] Nelson MB, Gilbert ON, Duncan PW, Kitzman DW, Reeves GR, Whellan DJ, Mentz RJ, Chen H, Hewston LA, Taylor KM, Pastva AM. Intervention Adherence in REHAB-HF: Predictors and Relationship With Physical Function, Quality of Life, and Clinical Events. J Am Heart Assoc. 2022 Jun 7;11(11):e024246. doi: 10.1161/JAHA.121.024246. Epub 2022 Jun 3. PMID 35656973
- [Derived] Mentz RJ, Whellan DJ, Reeves GR, Pastva AM, Duncan P, Upadhya B, Nelson MB, Chen H, Reed SD, Rosenberg PB, Bertoni AG, O'Connor CM, Kitzman DW. Rehabilitation Intervention in Older Patients With Acute Heart Failure With Preserved Versus Reduced Ejection Fraction. JACC Heart Fail. 2021 Oct;9(10):747-757. doi: 10.1016/j.jchf.2021.05.007. Epub 2021 Jul 7. PMID 34246602
- [Derived] Kitzman DW, Whellan DJ, Duncan P, Pastva AM, Mentz RJ, Reeves GR, Nelson MB, Chen H, Upadhya B, Reed SD, Espeland MA, Hewston L, O'Connor CM. Physical Rehabilitation for Older Patients Hospitalized for Heart Failure. N Engl J Med. 2021 Jul 15;385(3):203-216. doi: 10.1056/NEJMoa2026141. Epub 2021 May 16. PMID 33999544
- [Derived] Warraich HJ, Kitzman DW, Whellan DJ, Duncan PW, Mentz RJ, Pastva AM, Nelson MB, Upadhya B, Reeves GR. Physical Function, Frailty, Cognition, Depression, and Quality of Life in Hospitalized Adults >/=60 Years With Acute Decompensated Heart Failure With Preserved Versus Reduced Ejection Fraction. Circ Heart Fail. 2018 Nov;11(11):e005254. doi: 10.1161/CIRCHEARTFAILURE.118.005254. PMID 30571197
- [Derived] Reeves GR, Whellan DJ, O'Connor CM, Duncan P, Eggebeen JD, Morgan TM, Hewston LA, Pastva A, Patel MJ, Kitzman DW. A Novel Rehabilitation Intervention for Older Patients With Acute Decompensated Heart Failure: The REHAB-HF Pilot Study. JACC Heart Fail. 2017 May;5(5):359-366. doi: 10.1016/j.jchf.2016.12.019. Epub 2017 Mar 8. PMID 28285121

RESULTS

PARTICIPANT FLOW:
Groups:
- Attention Control: Usual care group with bi-weekly contact
- Rehabilitation Intervention: Individual, tailored, progressive, multi-domain physical function rehabilitation intervention
Period: Overall Study
Arm/Group | Attention Control | Rehabilitation Intervention
Started | 174 | 175
Completed | 157 | 153
Not Completed | 17 | 22
Not completed — Death | 16 | 21
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Attention Control | Rehabilitation Intervention | Total
Number analyzed (Participants) | 174 | 175 | 349
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.2 (7.7) | 73.1 (8.5) | 72.7 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 85 | 183
  Male | 76 | 90 | 166
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 170 | 172 | 342
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 4 | 7
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 81 | 73 | 154
  White | 83 | 90 | 173
  More than one race | 5 | 6 | 11
  Unknown or Not Reported | 0 | 0 | 0
Short Physical Performance Battery [Mean (Standard Deviation); unit: Score on a Scale] — The Short Physical Performance Battery is scored on a scale of 0-12, with a higher score indicating better physical function.
  Score on a Scale | 6.1 (2.6) | 6.0 (2.8) | 6.1 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Short Physical Performance Battery (SPPB) at Month 3
Description: The Short Physical Performance Battery is scored on a scale of 0-12, with a higher score indicating better physical function.
Time Frame: Month 3
Population: Analysis completed on all participants alive with Month 3 SPPB obtained (n=304).
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Attention Control | Rehabilitation Intervention
Number analyzed (Participants) | 155 | 149
score on a scale | 6.9 (0.2) | 8.3 (0.2)
Statistical Analysis 1: Comparison: Attention Control vs Rehabilitation Intervention; Test type: Superiority; p < 0.0001, joint model; Joint model of ANCOVA plus survival; Mean Difference (Final Values) = 1.5, 95% CI 2-sided [0.9 to 2.0]

2. Secondary Outcome: All-Cause Rehospitalization
Description: Number of all-cause rehospitalizations 6 months from index hospital discharge.
Time Frame: Month 6
Population: All participants, regardless of participation in the intervention or Month 3 follow-up were followed for all-cause rehospitalizations. Analysis completed on all participants, including deaths, except participants lost to follow-up (n=1) and participants withdrawn from study (n=1).
Measure: Number; unit: rehospitalizations
Arm/Group | Attention Control | Rehabilitation Intervention
Number analyzed (Participants) | 173 | 174
rehospitalizations | 213 | 194
Statistical Analysis 1: Comparison: Attention Control vs Rehabilitation Intervention; Test type: Superiority; p = 0.59, Joint Model; Joint model of Poisson regression and survival; Rate Ratio = 0.93, 95% CI 2-sided [0.66 to 1.19]

3. Other Pre Specified Outcome: 6-minute Walk Distance
Description: Exploratory outcome. Distance walked in 6 minutes.
Time Frame: Month 3
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Handgrip Strength
Description: Exploratory outcome. Handgrip strength is measured in kilograms by a handgrip dynamometer.
Time Frame: Month 3
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Frailty Status (Fried Frailty Criteria) at Month 3
Description: Exploratory outcome. Frailty is assessed by the Fried criteria consisting of 5 components: low physical activity, exhaustion, weakness, slowness, and unintentional weight loss. Presence of 3 or more Fried criteria indicates frailty, 1-2 criteria indicates pre-frailty, and 0 criteria indicates no frailty.
Time Frame: Month 3
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Quality of Life Measured by Kansas City Cardiomyopathy Questionnaire (KCCQ) Overall Summary Score
Description: Exploratory outcome. The KCCQ Overall Summary Summary Score is a heart failure disease-specific quality of life measure encompassing domains of physical limitation, HF symptoms, quality of life, and social limitation scored on a scale of 0-100 with higher scores indicating better health status.
Time Frame: Month 3
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Physical Limitation as Assessed by the KCCQ Physical Limitation Score
Description: Exploratory outcome. The Physical Limitation Score of the KCCQ questionnaire is a subscore evaluating disease-specific physical limitation. Scores range 0-100 with a higher score indicating less physical limitation.
Time Frame: Month 3
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Quality of Life Measured by Short Form 12 Item Questionnaire (SF-12)
Description: Exploratory outcome. The SF-12 is a quality of life assessment with 2 component scores (Physical Composite Score and Mental Composite Score) ranging 0-100 with higher scores indicating better health status.
Time Frame: Month 3
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Quality of Life Assessed by the EuroQol 5-dimension 5-level (EQ-5D-5L)
Description: Exploratory outcome. The EQ-5D-5L is a quality of life tool with 5 components designed to detect health utilities: mobility, usual activities, self-care, pain/discomfort, and anxiety/depression. All components are rated on a scale of 1-5 with higher scores indicating worse health status.
Time Frame: Month 6
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Depression Measured by the Geriatric Depression Scale
Description: Exploratory outcome. The Geriatric Depression Scale is a 15-item questionnaire evaluating depressive symptoms. Scores range from 0-15 with a higher score indicating more severe depressive symptoms.
Time Frame: Month 3
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Cognitive Function Measured by the Montreal Cognitive Assessment (MoCA)
Description: Exploratory outcome. The Montreal Cognitive Assessment is a tool for assessing multiple domains of cognitive function. Scores range 0-30 with higher scores indicating better cognitive function. A score greater than or equal to 26 is considered normal cognitive function.
Time Frame: Month 3
Reporting Status: Not Posted

12. Other Pre Specified Outcome: All-cause Rehospitalizations at Month 1
Description: Exploratory outcome. Number of all-cause rehospitalizations 1 month post index hospitalization discharge.
Time Frame: Month 1
Reporting Status: Not Posted

13. Other Pre Specified Outcome: All-cause Rehospitalizations at Month 3
Description: Exploratory outcome. Number of all-cause rehospitalizations 3 months after discharged from index hospitalization
Time Frame: Month 3
Reporting Status: Not Posted

14. Other Pre Specified Outcome: All-cause Combined Rehospitalization and Death at Month 6
Description: Exploratory outcome. Combined number of all-cause rehospitalizations and death 6 months after discharge from index hospitalization
Time Frame: Month 6
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Heart Failure Rehospitalizations at Month 6
Description: Exploratory outcome. Number of heart failure rehospitalizations 6 months after discharge from index hospitalization
Time Frame: Month 6
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Hospitalization Days Post-randomization
Description: Exploratory outcome. Total days spent hospitalized after date of randomization.
Time Frame: Month 6
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Facility-free Days Alive
Description: Exploratory outcomes. Total days alive spent outside of hospital, observation unit, acute rehab setting, and skilled nursing facility 6 months after discharge from index hospitalization.
Time Frame: Month 6
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Emergency Department Visits
Description: Exploratory outcomes. Number of emergency department visits after 6 months from hospital discharge
Time Frame: Month 6
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Observation Unit Stays <24 Hours
Description: Exploratory outcome. Number of observation unit stays <24 hours 6 months after discharge from index hospitalization
Time Frame: Month 6
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Unscheduled Urgent Medical Visits
Description: Exploratory outcome. Number of unscheduled urgent medical visits after discharge from index hospitalization
Time Frame: Month 6
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Global Rank Score of Short Physical Performance Battery Score + All-cause Rehospitalization + Death
Description: Exploratory outcome. The global rank composite outcome combines non-commensurate endpoints including death, number of all-cause rehospitalizations, and month 3 SPPB into a single non-parametric outcome in a hierarchical manner with death being ranked first and SPPB being ranked last. Participants are ranked from the most adverse response (lowest rank) to the most favorable response (highest rank).
Time Frame: Month 6
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Placement at Skilled Nursing Facility
Description: Exploratory outcome. Number of placements at skilled nursing facilities after discharge from index hospitalization.
Time Frame: Month 6
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Physical Activity Assessed by Accelerometry
Description: Exploratory outcome. Physical activity assessed by accelerometry quantified in moderate-vigorous physical activity minutes per day.
Time Frame: Month 6
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Generalized Optimism Assessed by the Life Orientation Test-Revised
Description: Exploratory outcome. The Life Orientation Test-Revised is a assessment of generalized optimism scored on a scale of 0-24 with higher scores indicating higher optimism.
Time Frame: Month 3
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Economic Analysis
Description: Assess direct medical costs, direct non-medical costs, indirect patient time costs, short-term cost-analysis, long-term cost analysis, and sustainability of the intervention.
Time Frame: Month 6
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Biomarkers
Description: Two well-accepted biomarkers of HF disease severity and prognosis, NT-proBNP and galectin-3, and increased biomarkers in older HF patients Tumor necrosis factor alpha, C-reactive protein, and interleukin-6.
Time Frame: Month 3
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: AEs collected from date of discharge from index hospitalization through Month 6.
Arm/Group | Attention Control | Rehabilitation Intervention
All-Cause Mortality (participants affected / at risk) | 16/174 | 21/175
Serious Adverse Events (participants affected / at risk) | 115/174 | 106/175
Other Adverse Events (participants affected / at risk) | 69/174 | 60/175
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Attention Control (N=174) | Rehabilitation Intervention (N=175)
anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
epitaxis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
aortic valve disease (Cardiac disorders) | 0 (0) | 1 (2)
atrial fibrillation (Cardiac disorders) | 1 (1) | 5 (5)
atrial flutter (Cardiac disorders) | 2 (2) | 2 (2)
bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
chest pain (Cardiac disorders) | 2 (3) | 6 (7)
heart failure exacerbation (Cardiac disorders) | 64 (107) | 57 (99)
mitral stenosis (Cardiac disorders) | 0 (0) | 2 (2)
mitral valve repair (Cardiac disorders) | 1 (1) | 1 (1)
myocardial infarction (Cardiac disorders) | 4 (5) | 2 (2)
sudden cardiac death (Cardiac disorders) | 1 (1) | 4 (4)
supraventricular tachycardia (Cardiac disorders) | 5 (5) | 4 (4)
ventricular tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
colitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
colonic fistula (Gastrointestinal disorders) | 0 (0) | 1 (2)
constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (2)
duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
gastroenteritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
gastrointestinal bleed (Gastrointestinal disorders) | 5 (5) | 4 (4)
gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
multiple organ failure (Gastrointestinal disorders) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 0 (0) | 1 (2)
small bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
edema (General disorders) | 1 (1) | 2 (2)
non-cardiac chest pain (General disorders) | 6 (6) | 6 (8)
cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 0 (0)
liver cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
primary amyloidosis (Immune system disorders) | 0 (0) | 1 (1)
bacterial endocarditis (Infections and infestations) | 0 (0) | 1 (1)
influenza (Infections and infestations) | 1 (1) | 0 (0)
osteomyelitis (Infections and infestations) | 2 (2) | 1 (1)
sepsis (Infections and infestations) | 2 (2) | 1 (1)
upper respiratory infection (Infections and infestations) | 2 (2) | 0 (0)
urinary tract infection (Infections and infestations) | 1 (1) | 2 (3)
wound infection (Infections and infestations) | 1 (1) | 0 (0)
fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
injurious fall (Injury, poisoning and procedural complications) | 16 (18) | 9 (10)
intracranial hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
oxycontin overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
serotonin syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
tacrolimus toxicity (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 1 (2) | 3 (3)
hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
gout flare (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
chronic lymphocytic leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
metastatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 2 (2)
pancreatic adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
dysarthia (Nervous system disorders) | 0 (0) | 1 (1)
neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
stroke (Nervous system disorders) | 4 (4) | 5 (6)
syncope (Nervous system disorders) | 3 (3) | 2 (3)
transient ischemic attack (Nervous system disorders) | 1 (1) | 0 (0)
sucidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
acute kidney injury (Renal and urinary disorders) | 6 (8) | 3 (3)
hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (3)
interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (3)
diabetic foot ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ablation (Surgical and medical procedures) | 2 (2) | 0 (0)
arteriovenous fistula placement (Surgical and medical procedures) | 0 (0) | 1 (1)
bronchoscopy (Surgical and medical procedures) | 0 (0) | 1 (1)
cateract surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
implantable cardioverter defibrillator implantation (Surgical and medical procedures) | 6 (7) | 1 (1)
pacemaker implantation (Surgical and medical procedures) | 0 (0) | 2 (2)
remodulin pump implantation (Surgical and medical procedures) | 0 (0) | 1 (1)
renal artery angioplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
hematoma (Vascular disorders) | 0 (0) | 1 (2)
hypertension (Vascular disorders) | 2 (2) | 1 (1)
hypotension (Vascular disorders) | 4 (4) | 2 (2)
pulmonary embolism (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Attention Control (N=174) | Rehabilitation Intervention (N=175)
anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
elevated international normalized ratio (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
epitaxis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
bradycardia (Cardiac disorders) | 0 (0) | 2 (2)
chest pain (Cardiac disorders) | 0 (0) | 2 (2)
heart failure exacerbation (Cardiac disorders) | 7 (7) | 7 (8)
suprventricular tachycardia (Cardiac disorders) | 0 (0) | 3 (3)
sudden vision loss (Eye disorders) | 0 (0) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
gastrointestinal pain (Gastrointestinal disorders) | 3 (3) | 2 (2)
melena (Gastrointestinal disorders) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
edema (General disorders) | 1 (1) | 0 (0)
fatigue (General disorders) | 0 (0) | 3 (3)
non-cardiac chest pain (General disorders) | 4 (4) | 5 (5)
weakness (General disorders) | 1 (1) | 0 (0)
upper respiratory infection (Infections and infestations) | 4 (4) | 4 (4)
urinary tract infection (Infections and infestations) | 1 (1) | 3 (4)
abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ear injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
fall (self-reported) (Injury, poisoning and procedural complications) | 62 (112) | 48 (94)
foot wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ICD device complications (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
inguinal hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
post-prodecural complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
fluid retention (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 4 (5)
hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
gout flare (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
muscle strain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 10 (13)
altered mental status (Nervous system disorders) | 0 (0) | 2 (2)
dizziness (Nervous system disorders) | 2 (2) | 8 (10)
headache (Nervous system disorders) | 0 (0) | 2 (2)
neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
seizure (Nervous system disorders) | 1 (1) | 0 (0)
syncope (Nervous system disorders) | 0 (0) | 1 (1)
acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
elevated creatinine (Renal and urinary disorders) | 0 (0) | 1 (1)
hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
kidney stone (Renal and urinary disorders) | 1 (1) | 1 (1)
urinary retention (Renal and urinary disorders) | 2 (2) | 0 (0)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
hypertension (Vascular disorders) | 0 (0) | 3 (4)
hypotension (Vascular disorders) | 0 (0) | 2 (2)
venous stasis (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-02-06): https://cdn.clinicaltrials.gov/large-docs/38/NCT02196038/Prot_SAP_000.pdf
  • Informed Consent Form (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/38/NCT02196038/ICF_001.pdf